CLINICAL TRIAL: NCT06079242
Title: Observational Study for SIR-Spheres Therapy for the Treatment of Unresectable Metastatic Liver Tumors From Primary Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: GrandPharma (China) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ST-GPL00102-CP001
Record Dates: First submitted 2023-09-22; First posted 2023-10-12 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Neoplasms
Keywords: Metastatic Colorectal Cancer; 90Y; Liver Metastases; SIRT; Radioembolization; SIR-Spheres Microspheres
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Resin microspheres containing yttrium-90 (Y-90) — SIR-Spheres Y-90 resin microspheres are permanent implant and for single use only
  Other Names: SIR-Spheres® Y-90

SUMMARY:
This real-world study tries to collect data reflecting routine use of SIR-Spheres in patients diagnosed with unresectable liver metastases from Metastatic Liver Tumors From Primary Colorectal Cancer (mCRC) refractory to or intolerant to chemotherapy, in order to assess clinical response in a real-world setting and further validate the safe and appropriate use of SIR-Spheres in China.

DETAILED DESCRIPTION:
This is a post-market trial evaluating the efficacy and safety of SIR-Spheres® Y-90 resin microspheres for the treatment of unresectable metastatic liver tumors from primary colorectal cancer. Patients enrolled should already complete the infusion of SIR-Spheres® and data are about to be collected both retrospectively and prospectively. 200 patients are anticipated to be enrolled and followed up for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Obtained informed consent for patients to be follow-up prospectively
2. Age≥18 years old
3. Histologically or pathologically confirmed diagnosis of unresectable metastatic liver tumors from primary colorectal cancer and failed standard of care
4. Received SIR-Spheres®

Exclusion Criteria:

1. Special contraindications from package insert, which includes

   1. Markedly abnormal liver function tests, such as total bilirubin > 2.0 mg/dL or albumin <3.0 g/dL
   2. Portal vein thrombosis in the main trunk
   3. Disseminated extrahepatic disease
   4. Previous external beam radiation therapy to the liver
2. Women are lactating or pregnant during the study or plan to be pregnant during the study
3. Patients with mental illness or cognitive impairment
4. Per investigator, patients are non-adherent or reluctant to be followed up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresectable metastatic liver tumors from primary colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Liver-specific overall response rate (ORR) according to RECIST 1.1 | 24 months
  Percentage of subjects with complete or partial responses to the liver as determined by the investigator according to liver-specific RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall survival (OS) | 24 months
  From the day of treatment with yttrium [90Y] resin microspheres to the time of death due to any cause
1-yr OS | 12 months
  The percentage of subjects treated with yttrium [90Y] resin microspheres who survived at 1 year.
Progression-free survival(PFS) assessed by the investigator | 24 months
  Defined as the time from the date of treatment with the yttrium [90Y] resin microspheres to the time when disease progression or subject death from any cause during the study period was first determined by the investigator according to RECIST 1.1 criteria, whichever occurred first.
Liver-specific PFS assessed by the investigator | 24 months
  Defined as the time from the date of treatment with yttrium [90Y] resin microspheres until the first time progression of liver disease or death of the subject from any cause during the study period was determined by the investigator according to liver-specific RECIST 1.1 criteria, whichever occurred first.
ORR assessed by the investigator | 24 months
  Defined as the percentage of subjects with complete or partial tumor response as determined by the investigator according to RECIST 1.1 criteria
Objective Duration of tumor response (DOR) assessed by the investigator | 24 months
  Defined as the time from the first documented objective response to tumor recurrence or death from any cause during the study period as determined by the investigator according to RECIST 1.1 criteria, whichever occurs first
Duration of liver-specific DOR assessed by the investigator | 24 months
  Defined as the time from the first documented liver objective remission to liver recurrence or death from any cause during the study period as determined by the investigator according to liver-specific RECIST 1.1 criteria, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided